CLINICAL TRIAL: NCT02349802
Title: Evaluation of the Single-Use Pre-Filled Autoinjector
Brief Title: Autoinjector Device Assessment Study
Acronym: BCB119
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5554C00001
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Subjects
Keywords: Auto-injector Device, device-related injection, Auto-injector
MeSH Terms: interventions — Syringes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Experimental): exenatide suspension - 9 mg / 0.85 mL
  Interventions: Drug: Auto-injector with exenatide suspension
- Arm 2 (Experimental): exenatide suspension - 9 mg / 0.85 mL
  Interventions: Drug: Syringe with exenatide suspension
- Arm 3 (Experimental): exenatide suspension - 4.5 mg /1.1 mL
  Interventions: Drug: Syringe with exenatide suspension
- Arm 4 (Experimental): exenatide suspension - 9 mg / 1.1 mL
  Interventions: Drug: Syringe with exenatide suspension
- Arm 5 (Experimental): exenatide suspension - 9 mg / 1.5 mL
  Interventions: Drug: Syringe with exenatide suspension

INTERVENTIONS:
Drug: Auto-injector with exenatide suspension — A flexible study design to accommodate multiple cohorts.
  Arms: Arm 1
Drug: Syringe with exenatide suspension — A flexible study design to accommodate multiple cohorts.
  Arms: Arm 2; Arm 3; Arm 4; Arm 5

SUMMARY:
Phase I study to determine the device-related injection failure rate of the single-use, pre-filled autoinjector.

DETAILED DESCRIPTION:
Phase I multi-cohort study will employ a flexible study design to accommodate multiple cohorts. Healthy male or female subjects >or= 18 years with no significant health issues will be included. Each cohort will employ an open-label, single-arm, repeat-dose design. Injection failure rates will be continually assessed. Injection pain will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years old at Visit 1 (Screening). Subjects must be of legal age of consent.
* Has no significant health issues that would preclude study participation, as determined by medical history and physical examination
* Has body mass index of 22 kg/m2 to 45 kg/m2, inclusive, at Visit 1 (Screening)
* Has normal renal function (creatinine clearance adjusted for body surface area ≥90 mL/min/1.73 m2 as calculated using the MDRD equation) at Visit 1 (Screening)
* Is male, or is female and meets all the following criteria:

  1. Not breastfeeding
  2. Negative pregnancy test result (human chorionic gonadotropin, beta subunit [bhCG]) at Visit 1 (Screening)
  3. If of childbearing potential (including perimenopausal women who have had a menstrual period within 1 year), must practice and be willing to continue to practice appropriate birth control (defined as a method which results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as implants, injectables, hormonal contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation or occlusion, or a vasectomized partner) during the entire duration of the study. Subjects must practice appropriate birth control as stated above for 10 weeks after the last dose of study drug.
* Has no clinically significant abnormal laboratory test values (clinical chemistry, hematology, urinalysis) as judged by the investigator at Visit 1 (Screening)
* Has a physical examination and electrocardiogram (ECG) with no clinically significant abnormality, as judged by the investigator, at Screening
* Is able to read, understand, and sign the Informed Consent Forms (ICFs) and, if applicable, an Authorization to Use and Disclose Protected Health Information form (consistent with Health Insurance Portability and Accountability Act of 1996 [HIPAA] legislation), communicate with the investigator, and understand and comply with protocol requirements

Exclusion Criteria:

* Has a clinically significant medical condition that could potentially affect study participation and/or personal well-being, as judged by the investigator, including but not limited to the following conditions:

  1. History of, or currently have, acute or chronic pancreatitis, or have triglyceride concentrations

     * 500 mg/dL at Visit 1 (Screening)
  2. Presence of medullary carcinoma or multiple endocrine neoplasia (MEN II) OR a family history of medullary carcinoma or MEN II
  3. Organ transplantation
  4. Active cardiovascular disease within 3 months of Visit 1 such as myocardial infarction, clinically significant arrhythmia, unstable angina, coronary artery bypass surgery, or angioplasty; or are expected to require coronary artery bypass surgery or angioplasty during the course of the study. Subjects with stable cardiac disease are not excluded.
  5. Presence or history of severe congestive heart failure (New York Heart Association Class IV [CCNYHA 1994])
  6. Central nervous system disease, including epilepsy (individuals with a history of convulsions associated with hypoglycemia will not be excluded)
  7. Liver disease, acute or chronic hepatitis, alanine aminotransaminase (ALT), or serum glutamic pyruvic transaminase (SGPT) greater than 3 times the upper limit of the reference range
  8. History or presence of inflammatory bowel disease or other severe gastrointestinal diseases, particularly those which may impact gastric emptying, such as gastroparesis, pyloric stenosis, gastric bypass surgery or gastric banding surgery
  9. Clinically significant malignant disease (with the exception of basal and squamous cell carcinoma of the skin) within 5 years of Visit 1 (Screening)
  10. Hemoglobinopathy, hemolytic anemia, or anemia (hemoglobin concentration below the lower limit of normal unless deemed not clinically significant by the investigator)
  11. Two or more episodes of severe hypoglycemia within 6 months prior to Visit 1. Refer to Section 9.1.5.2 for more information on hypoglycemia
  12. Evidence of acute or chronic illness including known or suspected human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) infection
* Has any abdominal skin abnormalities (e.g., extensive scarring, burns, inflammation, hyperkeratosis, etc.) which, in the investigator's opinion, could interfere with the injection.
* Has serum calcitonin concentration ≥100 pg/mL at Visit 1 (Screening)
* Has evidence of current abuse of drugs or alcohol or a history of abuse that, in the investigator's opinion, would cause the individual to be noncompliant
* Has a positive urine drug screen (including screen for cocaine, opiates, amphetamines, and cannabinoids)
* Has received any investigational drug within 30 days (or 5 half-lives of the investigational drug, whichever is greater) prior to Visit 1 (Screening)
* Has donated blood or had a significant blood loss within 2 months of first dose of study drug or is planning to donate blood during the study
* Has had a major surgery or a blood transfusion within 2 months prior to Visit 1 (Screening)
* Has known contraindication, allergies, or hypersensitivity to any component of study drug (including poly-D,L lactide co-glycolide [PLG] and MCT)
* Is employed by Amylin, Alkermes, Bristol-Myers Squibb, or AstraZeneca (i.e. that is an employee, temporary contract worker, or designee responsible for the conduct of the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3052 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of device-related failure injections | 10 week study
  The primary outcome measure is the number of device-related injection failures of the single-use, pre-filled auto-injector.

SECONDARY OUTCOMES:
Number of device-related injection failures of alternate device configuration | 10 week study
  The secondary outcome measure is the number of device-related injection failures of alternate device configuration.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, MD, Principal Investigator — Celerion; Peter Davidson, DO, Principal Investigator — Celerion; Elise Hardy, MD, Study Director — AstraZeneca
Locations (2):
- United States (2):
  - Research Site, Tempe, Arizona
  - Research Site, Lincoln, Nebraska

REFERENCES:
- See also: D5554C00001_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2631&filename=D5554C00001_CSR_Synopsis.pdf